CLINICAL TRIAL: NCT04230486
Title: Virtual Reality System for Cross-modal Rehabilitation of Hemianopia
Brief Title: VR System for Cross-modal Rehabilitation of Hemianopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061542
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-02

CONDITIONS: Hemianopia, Homonymous; Hemianopsia, Homonymous
Keywords: Hemianopia; Virtual Reality; Rehabilitation; Hemianopsia
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Intervention Model Description: All study participants will be given the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Experimental Group Virtual Reality (VR) Treatment (Experimental): Visual Auditory Virtual Reality rehabilitation for visual hemianopia
  Interventions: Device: Cross-model Visual Auditory Rehabilitation

INTERVENTIONS:
Device: Cross-model Visual Auditory Rehabilitation — Subjects will put on a virtual reality rehabilitation system which will present sights and sounds.

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a new rehabilitation for visual hemianopia. The study team believes a cross-modal rehabilitation technique delivered by a virtual reality system can help restore the visual field for subjects with homonymous hemianopia.

DETAILED DESCRIPTION:
The study tests a novel rehabilitation system, translated from promising cross-modal rehabilitation animal research, that is the first treatment capable of restoring the visual field for hemianopia patients. This noninvasive technique uses a virtual reality device to deliver visual and auditory stimulus. The goals of this study are to obtain proof of concept and procure rehabilitation data to support the development of this novel rehabilitation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers diagnosed with homonymous visual hemianopia / hemianopsia (ages 18-99)

Exclusion Criteria:

* Volunteers who are unable to complete the study tasks or understand instructions
* Subjects that are not able to provide written consent or verbal assent
* Subjects who are not available to complete all rehabilitation sessions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huai Jiang, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that underlie the results reported in the publication will be shared after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available immediately following publication for five years.
Access Criteria: Anyone who wishes to access the data for any purpose.
URL: https://github.com/Huai-Jiang/VR-Rehab

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six subjects signed consent. One screen failed.
Period: Overall Study
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Started | 6
Completed | 5
Not Completed | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Population: Analysis population includes only subjects who met screening criteria.
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (13.667)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Humphrey Visual Field Perimetry
Description: The area of the subject's visual field measured by 30-2 Humphrey visual field (HVF) perimetry. Both left and right sides will be tested. The deficit side includes is the hemianopic side. The intact side is the non-hemianopic side. During the HVF test, light is projected into a white bowl with a standardized background light intensity to form a circular stimulus, around 30 cm away from the patient's eye. The overall field mapping technique used is a form of static perimetry, where a stimulus appears in various areas of the field of vision. The patient indicates when they can see the stimulus and the perimetrist then records the point where the stimulus was seen. These data points are used to determine the patient's visual field.
Time Frame: Baseline
Population: Analysis only includes subjects who completed study.
Measure: Mean (Standard Deviation); unit: visual angle degrees^2
Units Other Than Participants: eyes
Groups:
- Virtual Reality (VR) Treatment--Deficit Eye: Visual Auditory Virtual Reality rehabilitation for visual hemianopia group--deficit eye. Deficit eye is the hemianopic side.
- Virtual Reality (VR) Treatment-Intact: Visual Auditory Virtual Reality rehabilitation for visual hemianopia group--intact eye. Intact eye is non-hemianopic side.
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 5 | 5
Number analyzed (eyes) | 5 | 5
visual angle degrees^2 | 108 (198.49) | 1272 (117.58)

2. Primary Outcome: Humphrey Visual Field Perimetry
Description: as for outcome 1
Time Frame: up to 2 Months
Population: Analysis only includes subjects who completed study.
Measure: Mean (Standard Deviation); unit: visual angle degrees^2
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 5 | 5
Number analyzed (eyes) | 5 | 5
visual angle degrees^2 | 594 (542.99) | 1356 (18.59)

3. Primary Outcome: Virtual Reality (VR) Visual Field Test--Mean Percent Correct
Description: Percent of correct trials in each location tested. Location at 15 degrees and 30 degrees on the horizontal meridian on both the left and right side were tested. Virtual Reality Visual Field test is a brief 5-minute test using the VR system to track rehabilitation progress. The test consists of 30 trials with visual stimulus presented either 15° or 30° in either the hemianopia field or the intact field at random time intervals.
Time Frame: Day 1
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 0 (0) | 91.667 (11.785)
  30 Degrees | 8.33 (11.785) | 100 (0)

4. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 2
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 16.667 (23.57) | 100 (0)
  30 Degrees | 0 (0) | 100 (0)

5. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 3
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 8.333 (11.785) | 100 (0)
  30 Degrees | 0 (0) | 100 (0)

6. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 4
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 0 (0) | 100 (0)
  30 Degrees | 0 (0) | 100 (0)

7. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 5
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 0 (0) | 100 (0)
  30 Degrees | 8.333 (11.785) | 100 (0)

8. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 6
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 8.333 (11.785) | 100 (0)

9. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 7
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 58.333 (35.355) | 100 (0)
  30 Degrees | 8.333 (11.785) | 100 (0)

10. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 8
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19. One subject did not complete the test day 8, so no data was collected for any subjects for this day.
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 0 | 0
Number analyzed (eyes) | 0 | 0

11. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 9
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 8.333 (11.785) | 100 (0)

12. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 10
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 8.333 (11.785) | 100 (0)

13. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 11
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19. One subject did not complete the test day 11, so no data was collected for any subjects for this day.
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 0 | 0
Number analyzed (eyes) | 0 | 0

14. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 12
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 8.33 (11.785) | 91.667 (11.785)

15. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 13
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 41.667 (58.926) | 100 (0)
  30 Degrees | 8.333 (11.785) | 100 (0)

16. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 14
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 58.333 (58.926) | 100 (0)
  30 Degrees | 8.333 (11.785) | 100 (0)

17. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 15
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 91.667 (11.785)
  30 Degrees | 8.333 (11.785) | 100 (0)

18. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 16
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 0 (0) | 100 (0)

19. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 17
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 0 (0) | 100 (0)

20. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 18
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 0 (0) | 100 (0)

21. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 19
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 0 (0) | 91.667 (11.785)

22. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 20
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 8.333 (11.785) | 100 (0)

23. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 21
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19. One subject did not complete the test day 21, so no data was collected for any subjects for this day.
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 0 | 0
Number analyzed (eyes) | 0 | 0

24. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 22
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (47.14) | 100 (0)
  30 Degrees | 41.667 (58.926) | 91.667 (11.785)

25. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 23
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19. One subject did not complete the test day 23, so no data was collected for any subjects for this day.
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 0 | 0
Number analyzed (eyes) | 0 | 0

26. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 24
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19. One subject did not complete the test day 24, so no data was collected for any subjects for this day.
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 0 | 0
Number analyzed (eyes) | 0 | 0

27. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 25
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 66.667 (47.14) | 100 (0)
  30 Degrees | 58.333 (58.926) | 100 (0)

28. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 26
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 50 (70.711) | 100 (0)
  30 Degrees | 50 (70.711) | 100 (0)

29. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 27
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19. One subject did not complete the test day 27, so no data was collected for any subjects for this day.
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 0 | 0
Number analyzed (eyes) | 0 | 0

30. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 28
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19. Data was not collected for 3 subjects due to logistical issues during COVID-19. One subject did not complete the test day 28, so no data was collected for any subjects for this day.
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 0 | 0
Number analyzed (eyes) | 0 | 0

31. Primary Outcome: Virtual Reality Visual Field Test--Mean Percent Correct
Description: as for outcome 3
Time Frame: Day 29
Population: Data was not collected for 3 subjects due to logistical issues during COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 2 | 2
Number analyzed (eyes) | 2 | 2
percentage of correct trials
  15 Degrees | 66.667 (47.14) | 100 (0)
  30 Degrees | 50 (70.711) | 100 (0)

32. Primary Outcome: Peripheral Visual Field Frame Test
Description: The number of points subjects can detect in each location of the visual field along the horizontal meridian. Percent of correct trials in each location tested in the deficit and intact side. Locations at 15°, 30°, 45°, 60°, and 75° on the horizontal meridian on the left and right side were tested.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 5 | 5
Number analyzed (eyes) | 5 | 5
Percent of correct trials
  15 Degrees | 20 (44.7214) | 80 (44.7214)
  30 Degrees | 20 (44.7214) | 80 (44.7214)
  45 Degrees | 20 (44.7214) | 80 (44.7214)
  60 Degrees | 20 (44.7214) | 72 (43.8178)
  75 Degrees | 0 (0) | 76 (43.359)

33. Primary Outcome: Peripheral Visual Field Frame Test
Description: as for outcome 32
Time Frame: up to 2 Months
Measure: Mean (Standard Deviation); unit: Percent of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 5 | 5
Number analyzed (eyes) | 5 | 5
Percent of correct trials
  15 Degrees | 100 (0) | 80 (44.7214)
  30 Degrees | 96 (8.9443) | 96 (8.9443)
  45 Degrees | 92 (17.8885) | 100 (0)
  60 Degrees | 80 (44.7214) | 100 (0)
  75 Degrees | 60 (54.7723) | 92 (17.8885)

34. Primary Outcome: Peripheral Visual Field Frame Test
Description: as for outcome 32
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: Percent of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 5 | 5
Number analyzed (eyes) | 5 | 5
Percent of correct trials
  15 Degrees | 95 (10) | 90 (20)
  30 Degrees | 90 (20) | 90 (20)
  45 Degrees | 80 (40) | 100 (0)
  60 Degrees | 75 (50) | 100 (0)
  75 Degrees | 65 (47.2582) | 100 (0)

35. Primary Outcome: Peripheral Visual Field Frame Test
Description: as for outcome 32
Time Frame: 6 Months
Population: Due to study timeline constraints, only one subject completed the 6 month follow-up test.
Measure: Number; unit: Percent of correct trials
Units Other Than Participants: eyes
Arm/Group | Virtual Reality (VR) Treatment--Deficit Eye | Virtual Reality (VR) Treatment-Intact
Number analyzed (Participants) | 1 | 1
Number analyzed (eyes) | 1 | 1
Percent of correct trials
  15 Degrees | 100 | 100
  30 Degrees | 100 | 100
  45 Degrees | 100 | 100
  60 Degrees | 100 | 100
  75 Degrees | 100 | 100

36. Secondary Outcome: National Eye Institute Visual Function Questionnaire (NEI-VFQ-25)--Composite Score
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. This score is calculated from the average of all subscale scores in the NEI VFQ-25 excluding the general health score. The score ranges from 0 to 100. A higher score denotes better vision-related quality of life.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 60.793 (19.498)
  2 months | 68.621 (21.932)
  3 months | 69.893 (29.418)

37. Secondary Outcome: NEI-VFQ-25--Composite Score
Description: as for outcome 36
Time Frame: 6 month
Population: The study's start was delayed due to COVID so only 1 participant was able to complete the 6 month follow-up within the grant time frame.
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 85.87

38. Secondary Outcome: NEI-VFQ-25--General Health Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The General Health Score is a subscale that measures the participant's self-report of their overall health. The score ranges from 0 to 100. A higher score denotes better perception of overall health.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 68.75 (37.5)
  2 months | 68.75 (31.458)
  3 months | 62.5 (17.678)

39. Secondary Outcome: NEI-VFQ-25--General Health Score Subscale
Description: as for outcome 38
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 50

40. Secondary Outcome: NEI-VFQ-25--General Vision Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The General Vision Score measures the participant's reported quality of vision. The score ranges from 0 to 100. A higher score denotes a better perception of vision
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 65 (19.149)
  2 months | 60 (28.284)
  3 months | 70 (14.142)

41. Secondary Outcome: NEI-VFQ-25--General Vision Score Subscale
Description: as for outcome 40
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 80

42. Secondary Outcome: NEI-VFQ-25--Ocular Pain Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Ocular Pain Score Subscale measures reported pain or discomfort in and around the eyes. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life related to ocular pain.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 90.625 (6.25)
  2 months | 90.625 (11.968)
  3 months | 81.25 (26.517)

43. Secondary Outcome: NEI-VFQ-25--Ocular Pain Score Subscale
Description: as for outcome 42
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 100

44. Secondary Outcome: NEI-VFQ-25--Near Activities Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Near Activities Score Subscale measures difficulty with performing near activities. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life related to near activities.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 56.25 (22.948)
  2 months | 60.417 (31.458)
  3 months | 75 (11.785)

45. Secondary Outcome: NEI-VFQ-25--Near Activities Score Subscale
Description: as for outcome 44
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 75

46. Secondary Outcome: NEI-VFQ-25--Distance Activities Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Distance Activities Score Subscale measures difficulty with performing distance activities. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life related to distance activities.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 48.333 (18.609)
  2 months | 76.25 (19.167)
  3 months | 77.5 (20.035)

47. Secondary Outcome: NEI-VFQ-25--Distance Activities Score Subscale
Description: as for outcome 46
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 75

48. Secondary Outcome: NEI-VFQ-25--Social Functioning Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Social Functioning Score Subscale measures how vision difficulties affect social functioning. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life related to social functioning.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 55 (24.495)
  2 months | 70.625 (35.259)
  3 months | 87.5 (17.678)

49. Secondary Outcome: NEI-VFQ-25--Social Functioning Score Subscale
Description: as for outcome 48
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 87.5

50. Secondary Outcome: NEI-VFQ-25--Mental Health Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Mental Health Score Subscale measures how much patients feel vision affects their mental health. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life relating to mental health.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 51.563 (32.022)
  2 months | 48.4375 (35.858)
  3 months | 56.25 (61.872)

51. Secondary Outcome: NEI-VFQ-25--Mental Health Score Subscale
Description: as for outcome 50
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 98.73

52. Secondary Outcome: NEI-VFQ-25--Role Difficulties Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Role Difficulties Score Subscale measures how limited by their vision patients feel they are. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life relating to role difficulties.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 62.5 (32.275)
  2 months | 65.625 (11.968)
  3 months | 50 (70.711)

53. Secondary Outcome: NEI-VFQ-25--Role Difficulties Score Subscale
Description: as for outcome 52
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 100

54. Secondary Outcome: NEI-VFQ-25--Dependency Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Dependency Score Subscale measures how much patients are dependent on other people due to their vision. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life related to dependency.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 41.667 (35.355)
  2 months | 50 (41.388)
  3 months | 62.5 (53.033)

55. Secondary Outcome: NEI-VFQ-25--Dependency Score Subscale
Description: as for outcome 54
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 100

56. Secondary Outcome: NEI-VFQ-25--Driving Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Driving Score Subscale measures patients' reported difficulty with driving. The score ranges from 0 to 100. Patients who do not drive are not given a driving score. A higher score denotes better vision-specific quality of life related to driving.
Time Frame: Baseline, 2 months, 3 months
Population: Driving Score Mean and Standard deviation could not be calculated because only one subject was driving and only for the 3 month follow up.
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale
  Baseline: number analyzed (Participants) | 0
  2 months: number analyzed (Participants) | 0
  3 months | 83.333

57. Secondary Outcome: NEI-VFQ-25--Driving Score Subscale
Description: as for outcome 56
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 58.33

58. Secondary Outcome: NEI-VFQ-25--Color Vision Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Color Vision Score Subscale measures how much difficulty patients have with using color vision to complete daily activities such as picking out clothes. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life related to color vision.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 75 (20.412)
  2 months | 87.5 (14.434)
  3 months | 87.5 (17.678)

59. Secondary Outcome: NEI-VFQ-25--Color Vision Score Subscale
Description: as for outcome 58
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 100

60. Secondary Outcome: NEI-VFQ-25--Peripheral Vision Score Subscale
Description: The NEI-VFQ-25 is a 25-item questionnaire regarding the quality of vision, social functioning, visual dependency, near vision, and color vision. The Peripheral Vision Score Subscale measures how much difficulty patients have with their peripheral vision to complete daily activities. The score ranges from 0 to 100. A higher score denotes better vision-specific quality of life related to peripheral vision.
Time Frame: Baseline, 2 months, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 50 (35.3554)
  2 months | 81.25 (37.5)
  3 months | 62.5 (17.678)

61. Secondary Outcome: NEI-VFQ-25--Peripheral Vision Score Subscale
Description: as for outcome 60
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: score on a scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
score on a scale | 75

62. Secondary Outcome: Veterans Affairs Low Vision Visual Function Questionnaire-48 (VA LV VFQ-48)--Item Score
Description: The VA LV VFQ-48 is a self-report instrument designed to measure difficulty visually impaired persons have performing daily activities. The acceptable range for the average item score is <= 2.34 (most difficult) and >=-2.22 (least difficult). Scores out of this range indicate something other than visual impairment is governing the patient's responses. The Item Score is the average functional reserve of all the items in the questionnaire excluding items which were rated Unscored (Difficult / don't do for Non-Visual Reasons). Functional reserve is the difference between a patient's visual ability and the visual ability needed to perform an activity.
Time Frame: Baseline, 2 months
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
Score on a Scale
  Baseline | 1.248 (0.898)
  2 Months | 1.704 (0.948)

63. Secondary Outcome: VA LV VFQ-48--Item Score
Description: as for outcome 62
Time Frame: 3 months
Population: Only one subject completed this outcome measure during the 3 month follow-up due to study timeline constraints.
Measure: Number; unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
Score on a Scale | 2.063

64. Secondary Outcome: VA LV VFQ-48--Item Score
Description: as for outcome 62
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
Score on a Scale | 1.955

65. Secondary Outcome: VA LV VFQ-48--Composite Score
Description: The VA LV VFQ-48 is a self-report instrument designed to measure difficulty visually impaired persons have performing daily activities. The acceptable range for the average item score is <= 2.34 and >=-2.22. Scores out of this range indicate something other than visual impairment is governing the patient's responses. The reading domain score is calculated by calculating the average score of reading items. The composite score approximates a person's visual ability. The score is calculated using Massof's algorithm using the inverse hyperbolic tangent equation. For the composite score, a lower score is better.
Time Frame: Baseline, 2 months
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
Score on a Scale
  Baseline | -1.607 (1.923)
  2 Months | -2.481 (1.834)

66. Secondary Outcome: VA LV VFQ-48--Composite Score
Description: he VA LV VFQ-48 is a self-report instrument designed to measure difficulty visually impaired persons have performing daily activities. The acceptable range for the average item score is <= 2.34 and >=-2.22. Scores out of this range indicate something other than visual impairment is governing the patient's responses. The reading domain score is calculated by calculating the average score of reading items. The composite score approximates a person's visual ability. The score is calculated using Massof's algorithm using the inverse hyperbolic tangent equation. For the composite score, a lower score is better.
Time Frame: 3 months
Population: Only one subject completed this outcome measure during the 3 month follow-up due to study timeline constraints.
Measure: Number; unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
Score on a Scale | -2.415

67. Secondary Outcome: VA LV VFQ-48--Composite Score
Description: as for outcome 66
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
Score on a Scale | -2.095

68. Secondary Outcome: VA LV VFQ-48--Reading Domain Score
Description: The VA LV VFQ-48 is a self-report instrument designed to measure difficulty visually impaired persons have performing daily activities. The reading domain score is calculated by calculating the average score of reading items. Scores range from 0 to 3.5 logits, with higher scores denoting better ability to perform activities. The Reading Domain Score is the average functional reserve of the items measuring the reading functional domain, excluding items which were rated Unscored (Difficult / don't do for Non-Visual Reasons).
Time Frame: Baseline, 2 months
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 5
Score on a Scale
  Baseline | 1.839 (1.050)
  2 Months | 2.230 (0.982)

69. Secondary Outcome: VA LV VFQ-48--Reading Domain Score
Description: as for outcome 68
Time Frame: 3 months
Population: Only one subject completed this outcome measure during the 3 month follow-up due to study timeline constraints.
Measure: Number; unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
Score on a Scale | 2.673

70. Secondary Outcome: VA LV VFQ-48--Reading Domain Score
Description: as for outcome 68
Time Frame: 6 months
Population: as for outcome 37
Measure: Number; unit: Score on a Scale
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
Number analyzed (Participants) | 1
Score on a Scale | 2.549

71. Other Pre Specified Outcome: Grating Acuity Test
Description: Change in the percentage of correctly identified trials.
Time Frame: First visit after the completion of rehabilitation (1 or 2 months)
Reporting Status: Not Posted

72. Other Pre Specified Outcome: Color Vision Test
Description: Change in the percentage of correctly identified trials for each color.
Time Frame: First visit after the completion of rehabilitation (1 or 2 months)
Reporting Status: Not Posted

73. Other Pre Specified Outcome: Shape Recognition Test
Description: Change in the percentage of correctly identified trials.
Time Frame: First visit after the completion of rehabilitation (1 or 2 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through 6 months
Arm/Group | Experimental Group Virtual Reality (VR) Treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT04230486/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT04230486/ICF_000.pdf